CLINICAL TRIAL: NCT01728051
Title: An Open Label, Expanded Access Study of Melphalan Chemosaturation With the Delcath System in Patients With Ocular and Cutaneous Melanoma Metastatic to the Liver
Brief Title: Expanded Access Study of Melphalan With Delcath CS-PHP System in Patients With Ocular/Cutaneous Melanoma Mets to Liver
Status: No longer available | Type: Expanded Access
Sponsor: Delcath Systems Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MEL 2009-01
Record Dates: First submitted 2012-11-13; First posted 2012-11-16 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Metastatic Liver Cancer; Ocular Melanoma; Cutaneous Melanoma
MeSH Terms: conditions — Liver Neoplasms; Uveal Melanoma; Melanoma | interventions — Melphalan

INTERVENTIONS:
Drug: Melphalan
Device: Percutaneous Hepatic Perfusion

SUMMARY:
The safety and efficacy of CS-PHP-melphalan has been evaluated in a phase 3 trial conducted in the same patient population as well as using the same melphalan dosing as proposed in this study. This expanded access protocol will provide an experimental alternative treatment option for both physicians and patients until the Delcath CS-PHP System receives marketing approval.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven ocular/cutaneous melanoma with liver-dominant unresectable metastatic disease, defined as limited extra-hepatic disease and hepatic involvement which would, in the Investigator's opinion, result in morbidity and eventual mortality. Limited extra-hepatic disease considered acceptable includes:

   * up to 4 pulmonary nodules, each <1cm in diameter
   * retroperitoneal lymph nodes <1cm in diameter
   * resectable skin or subcutaneous metastases
   * asymptomatic bone metastases that have been, or can be, palliated with external beam radiation therapy
   * a solitary metastasis to any site that can be resected with limited morbidity or controlled with radiation
2. ≥1 measurable hepatic lesion per RECIST 1.1
3. Vasculature compatible with insertion of CS-PHP catheters, per baseline abdominal MRA
4. ECOG PS 0-2

Exclusion Criteria:

1. Chemotherapy, radiotherapy, or biologic therapy for the malignancy ≤1 month prior to 1st CS-PHP-melphalan infusion
2. Extensive prior radiotherapy, defined as treatment to ≥50% of marrow-containing bones
3. Immunosuppressive drugs such as cyclosporine, tacrolimus, azathioprine, or long-term oral glucocorticoids taken currently or ≤3 mths prior to 1st CS-PHP-melphalan infusion
4. Received an investigational product ≤30 days prior to the 1st CS-PHP-melphalan infusion
5. History of orthotopic liver transplantation, untreated gastrinoma (i.e. gastric acid hypersecretion) or prior Whipple procedure
6. Not recovered from side effects of prior therapy to ≤ Grade 1 NCI CTCAE 4.03
7. Child's B or C cirrhosis, or clinical evidence of portal hypertension
8. Patients with >50% of liver replaced by tumor, histologic evidence of hepatic dysfunction seen by laparoscopic liver biopsy
9. History or evidence of clinically significant cardiac disease such as symptomatic arrhythmia, angina/ischemia, coronary artery bypass graft surgery or percutaneous transluminal coronary angioplasty, uncontrolled atrial fibrillation, CHF with a left ventricular ejection fraction <40%, uncontrolled hypertension (SBP >190 mmHg or DBP >100 mmHg), HR outside normal range of 50-100 bpm for women and 45-100 bpm for men
10. History/evidence of clinically significant pulmonary or cardiac disease incompatible with fitness to undergo general anesthesia
11. Uncontrolled diabetes mellitus or hypo/hyperthyroidism
12. Active uncontrolled infection
13. History of bleeding disorders or known unresolved venous shunting
14. Requirement for ongoing chronic anticoagulation
15. Evidence of intracranial abnormalities resulting in risk for bleeding with anticoagulation
16. History of alcohol or drug abuse ≤6 mths
17. Other malignancy within 3 yrs before enrollment with the exception of curatively treated basal or squamous cell carcinoma of the skin, or curatively treated cervical, breast carcinoma in situ or prostate cancer
18. History of hypersensitivity to: melphalan or its components; iodine contrast that cannot be controlled by premedication with antihistamines and steroids; latex
19. Known hypersensitivity to heparin in the presence of heparin-induced thrombocytopenia antibodies
20. Inadequate hematological or renal function as indicated by any of the following:

    * Platelets <100,000/mm3
    * Hb ≤10 g/dL
    * Neutrophils <2,000/mm3
    * S Creat >1.5 mg/dL or measured creatinine clearance <60 mL/min/1.73 m2
21. Inadequate liver function as indicated by any of the following:

    * Tbili ≥3.0 mg/dL
    * INR >1.5
    * AST/ALT >5xULN
22. Pregnant or nursing
23. Positive pregnancy test in subjects of childbearing potential ≤7 days prior to first CS-PHP-melphalan infusion
24. Women who are pre-menopausal (i.e. have had a menstrual period ≤12 months) who are unwilling or unable to undergo hormonal suppression to avoid menstruation during treatment
25. Sexually active females of childbearing potential and sexually active males with partners of reproductive potential unwilling or unable to use contraception from screening until at least 30 days after last administration of CS-PHP-melphalan

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Nutting, DO, Principal Investigator — Sky Ridge Medical Center; Jonathan Zager, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institue at University of Southern Florida; Mark Faries, MD, Principal Investigator — Saint John's Cancer Institute; James F Pingpank, MD, Principal Investigator — Univeristy of Pittsburg Cancer Center; Eric D Whitman, MD, Principal Investigator — Carol G. Simon Cancer Center at Morristown Memorial Hospital; H. Richard Alexander, MD, Principal Investigator — University of Maryland, Baltimore
Locations (6):
- United States (6):
  - John Wayne Cancer Institute at Saint John's Health Center, Santa Monica, California
  - Sky Ridge Medical Center, Englewood, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - University of Pittsburg Cancer Institute, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Related Info — http://www.delcath.com